CLINICAL TRIAL: NCT06505538
Title: Nurse-Led Mobile App Effect on Symptom Management for Breast Cancer Patients After Surgery: A Quasi-Experimental Study
Brief Title: Nurse-Led Mobile App Effect on Symptom Management for Breast Cancer Patients After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Collaborators: Semahat Arsel Nursing Education, Practice and Research Center (SANERC) (Unknown)
Responsible Party: Principal Investigator, Aydanur Aydin, MSc, PhD, RN, Associate Professor, Gümüşhane Universıty
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GumushaneUni1
Record Dates: First submitted 2024-03-01; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Symptom Management; Breast Care Nurse; Mobile App; Mobile Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Device: NL-Mapp
- Control (No Intervention)

INTERVENTIONS:
Device: NL-Mapp — Mobile applicaiton
  Arms: Intervention

SUMMARY:
Background: The use of the Nurse-Led Mobile App (NL-Mapp) is a current and important option for educating patients about the symptoms that may arise from breast cancer surgery.

Introduction: Given the precise information and counseling services offered to breast cancer patients, NL-Mapp is considered an appropriate choice to support postoperative self-care.

Methods: This quasi-experimental study aimed to determine the impact of NL-Mapp on breast cancer patients after surgery. The study included 45 patients in the intervention group and 45 patients in the control group. First, NL-Mapp was developed by the research team. Patients were then taught how to use the app to manage their symptoms after breast cancer surgery, and online counseling was provided for patients' questions. The intervention started before surgery, and follow-up visits were made before discharge and in the first month.

ELIGIBILITY:
Inclusion Criteria:

* Speaking the national language,
* The presence of primary breast cancer,
* The utilization of a smartphone for a minimum of one year,
* An age of 20 years

Exclusion Criteria:

* An uncontrollable medical problem,
* Having speech problems,
* Having hearing problems,
* Vision impairment,
* A psychiatric diagnosis/ongoing treatment
* Previous treatment due to a different type of cancer
* Rheumatological diseases,
* Fractures,
* Health problems leading to joint limitation,
* Amputation

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Function of the affected arm | three months
  ASES Shoulder Rating Scale
Body image and sexual adjustment scale | three months
  Sexual Adjustment and Body Image Scale
Pain scale | three months
  Visual Analog Scale

SECONDARY OUTCOMES:
Quality of life scale | one year
  Functional Assessment of Cancer Therapy-Breast

CONTACTS AND LOCATIONS:
Locations (1):
- Gumushane University, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aydin A, Gursoy A. Nurse-Led Mobile App Effect on Quality of Life in Breast Cancer Patients After Surgery: Nonrandomized Controlled Prospective Cohort Study (Step 3). Cancer Nurs. 2024 Nov 20. doi: 10.1097/NCC.0000000000001418. Online ahead of print. PMID 39565096